CLINICAL TRIAL: NCT06961682
Title: Effectiveness of MD on Patient With MetS to Control Hypertension, Diabetes ,Obesity and Dyslipidemia in Patients Attending Assiut University Hospital
Brief Title: Effectiveness of MD on MetS Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Gaber Osman, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Fam Med Dep AssiutU
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic syndrome patients attending Assiut university hospital (Experimental): MetS patients with diabetes, hypertension, dyslipidemia and obesity at least three criteria to diagnose the metabolic syndrome
  Interventions: Dietary Supplement: MD

INTERVENTIONS:
Dietary Supplement: MD — Red meats and sweets minimal consumption once or twice per month Eggs, cheese, poultry and yoghurt weekly consumption Fish and seafood two to three times per week Olive oil varing amount daily Vegetables and fruits daily consumption Legumes and whole grains (bread, pasta, rice and nuts )daily consumption Measure the effect of Mediterranean diet on patient with MetS to control hypertension, diabetes, obesity and dyslipidemia by measuring blood pressure mmHg regularly, Hba1c before, lipid profile LDL, HDL, TG weight (kg) and height (m) to calculate BMI wt kg/ht^2 m and waist hip ratio by measuring waist and hip circumference before and after the MD

SUMMARY:
The metabolic syndrome (MetS), is a complicated condition linked to coronary artery disease.This group includes visceral obesity (abdominal or android type obesity), insulin resistance (IR), hypertension, and dyslipidaemia.The global prevalence of MetS is estimated to be about one-quarter of the world population or over a billion global citizens .A high MetS prevalence of 55% was found in Egyptians, 85.6% among diabetics, and 76.6% among hypertensive patients .People can modify their diet, physical activity, decrease smoking habits to lower their chance of developing MetS. Frequent exercise can lower blood pressure while increasing insulin sensitivity, lipolysis, and energy expenditure. It has the ability to improve blood lipid parameters .Diet is one of the most important tools available to improve MetS. However, the diet for the prevention and treatment of MetS remains unspecified beyond weight control and reduction in total calories. Several evidences show that it should generally be low in saturated fats, trans fats, cholesterol, sodium and simple sugars .The adherence to the Mediterranean Diet(MD) brings up two positive features, firstly the activity levels are increased and secondly the environmental impact becomes self-rewarding. The more the MD is favoured, the more the self-productivity is achieved resulting in a stronger life style adaptation .MD causes reduction of CVD incidence and outcomes decreases BP (systolic and diastolic) , inverses association with mortality,improvements in dyslexia, decreases incidence of T2DM.

ELIGIBILITY:
1. Inclusion criteria:

   All people diagnosed as metabolic syndrome
   * (Hypertension(systolic BP≥130 or Diastolic BP ≥85)
   * prediabetes fasting plasma glucose(100-125),oral glucose tolerance test(140-199)Hba1c(5.7-6.4)ADA
   * Diabetes, fasting>125, oral glucose tolerance test>200, Hba1c≥6.5 ADA .
   * Hyperlipidaemia(TG≥150 mg\dl-HDL<40 in male and <50 in female) [12]
   * Obesity(waist circumference ≥102cm in male and ≥88cm in female) [12]
2. Exclusion criteria:

   * Type 1 diabetes
   * Patients with renal or advanced liver disease(Failure)
   * Oral contraceptives, psychiatric, neurologic medications and steroid therapy
   * Patients with heart failure and presence of stent
   * Endocrine disease (Thyroid disease especially hypothyroidism-Cushing disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessment the effectiveness of MD on obese MetS patients | 6 months
  by measuring weight in kg and height in meters to calculate BMI which equal weight\height square meters before and after MD at 3 and 6 months
Assessment the effectiveness of MD on hypertensive MetS patients | 6 months
  by regular measuring to blood pressure mmHg before and after the MD
Assessment the effectiveness of MD on diabetic MetS patients | 6 months
  by measuring Hga1c before and after the MD
Assessment the effectiveness of MD on dyslipidemic MetS patients | 6 months
  by measuring lipid profile HDL, LDL, TG

IPD SHARING:
Plan to Share IPD: No